CLINICAL TRIAL: NCT00863499
Title: International Study to Predict Optimised Treatment Response to Short or Long Acting Methylphenidate in Children and Adolescents With Attention Deficit/Hyperactivity Disorder.
Brief Title: International Study to Predict Optimised Treatment in Attention Deficit/Hyperactivity Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BRC Operations Pty. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: iSPOT-A
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Attention Deficit/Hyperactivity Disorder
Keywords: Attention Deficit/Hyperactivity Disorder; Attention Deficit Disorder; ADHD; ADD; iSPOT
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): Short Acting methylphenidate
  Interventions: Drug: Short Acting Methylphenidate
- B (Active Comparator): Long Acting Methylphenidate
  Interventions: Drug: Long Acting Methylphenidate
- C (No Intervention): Healthy Controls

INTERVENTIONS:
Drug: Short Acting Methylphenidate — Dosage: 5 mg twice daily (before breakfast and lunch) with gradual increments of 5 to 10 mg weekly. Daily dosage above 60 mg is not recommended.
  Other Names: • Ritalin; • Ritalina; • Attenta; • Methylin; • Penid; • Rubifen; *Consider treatment directions above or as physician directed as per usual care.
  Arms: A
Drug: Long Acting Methylphenidate — Dosage: 9 to 20 mg once daily in the morning (with or without food) with gradual increments of 9 to 20 mg weekly. Daily dosage above 60 mg is not recommended.
  Other Names: • Concerta; • Metadate CD; • Methylin ER; • Ritalin LA; • Ritalin Sustained-Release; *Consider treatment directions above or as physician directed as per usual care.
  Arms: B

SUMMARY:
The aim of the iSPOT-A study is to:

1. identify brain, genetic and cognitive markers of Attention Deficit/Hyperactivity Disorder, and
2. identify brain, genetic and cognitive markers that predict treatment response to short-acting methylphenidate in children and adolescents diagnosed with Attention Deficit/Hyperactivity Disorder.

DETAILED DESCRIPTION:
This is a multi-center, open-label effectiveness trial to identify objective indicators of treatment response in ADHD subjects (versus healthy controls) using cognitive and brain function measures, brain structure and genetic measures in subjects diagnosed with ADHD.

At least 672 naïve and treatment experienced subjects with ADHD will be enrolled from approximately 10 primary care centers. These patients are to be outpatients.

In addition, up to 672 healthy (non-ADHD) control subjects will be recruited who match the enrolled ADHD subjects in race, age, gender and years of education.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have signed an informed consent or assent form where required and/or whose parent or legal guardian has provided written informed consent.
* Subjects who meet DSM-IV criteria for primary diagnosis of ADHD at study entry, as determined by a psychiatrist, physician or clinical psychologist in conjunction with the clinical work-up undertaken by trained research assistants, as defined by The Mini International Neuropsychiatric Interview for Children and Adolescents (MINI Kid).
* Subjects who score at least 6 Inattentive or Hyperactive/impulsive items >1 on the Attention Deficit / Hyperactivity Disorder Rating Scale.
* Subjects who are stimulant naïve or stimulant free (defined as no stimulant medication in the previous 7 days*).
* Subjects who are 6-17 years of age (with an emphasis to enrol at least a third of the subjects who are ≥ 13 years of age).
* Subjects who are fluent and literate in English (and/or Dutch in The Netherlands).

  * coming off the stimulant medication for 7 days may place the participant at increased risk, therefore, the participant may have this washout period reduced to that defined in the drug package insert or 5 times the medication half life.

Exclusion Criteria:

* Known contra-indication or intolerance to the use of methylphenidate as defined in the product package insert (including previous treatment failure at the highest recommended dose).
* Pregnancy and females of child bearing potential who are not using a form of contraception and are at risk of becoming pregnant during the study.
* Known medical condition, disease or neurological disorder which might, in the opinion of investigator/s, interfere with the assessments to be made in the study or put ADHD patients at increased risk when exposed to optimal doses of the drug treatment. For example, a diagnosis of epilepsy would exclude a patient from this trial.
* History of physical brain injury or blow to the head that resulted in loss of consciousness for at least 10 minutes or at least 5minutes within the last two years. Prior treatment with methylphenidate or any other stimulant medication in the past 7 days.
* Known past or present substance dependence, including alcohol, as determined by The Mini International Neuropsychiatric Interview for Children and Adolescents (MINI Kid).
* Participation in an investigational study within four months of the baseline visit in which subjects have received an experimental drug/device that could affect the primary end points of this study.
* Use of any psychological or counselling therapy or CNS medication that cannot be washed out prior to participation or use of any psychological or counselling therapy between the baseline and week 6 (or Early Termination) visits.
* Subjects who, in the opinion of the investigator, have a severe impediment to vision, hearing and/or hand movement, which is likely to interfere with their ability to complete the testing batteries.
* Subjects who, in the opinion of the investigator, are unable and/or unlikely to comprehend and follow the study procedures and instructions.
* Presence of any other co-morbid primary DSM IV disorder.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1344 (Estimated)
Dates: Start 2009-10; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
To determine whether the genetic-brain-cognition function markers (or combination of markers) 'normalize' with acute drug treatment in ADHD. | 6 weeks

SECONDARY OUTCOMES:
To determine whether markers of acute treatment prediction are also predictive of functional outcome over 6-12 months. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A. Cohen, PhD, Principal Investigator — Center for Healing the Human Spirit; Harbans Multani, MD, Principal Investigator — Shanti Clinical Trials; Kamran Fallahpour, PhD, Principal Investigator — Brain Resource Center NY; Martijn Arns, PhD, Principal Investigator — Brainclinics Diagnostics B.V.; Mona Ismail, MD, Principal Investigator — Brain Resource Center NJ; Roger deBeus, PhD, Principal Investigator — Skyland Behavioral Health Associates; Simon Clarke, MD, Principal Investigator — Brain Dynamics Centre
Locations (7):
- United States (5):
  - Shanti Clinical Trials, Colton, California
  - Center for Healing the Human Spirit, Tarzana, California
  - Brain Resource Center, Englewood Cliffs, New Jersey
  - Brain Resource Center, New York, New York
  - Skyland Behavioral Health Associates , P.A., Asheville, North Carolina
- Brain Dynamics Centre, Westmead, New South Wales, Australia
- Brainclinics Diagnostics B.V., Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Leikauf JE, Griffiths KR, Clarke SD, Kohn MR, Williams L. Attention-Deficit/Hyperactivity Disorder Subtypes Defined by Cognition Have a Distinct Neural and Clinical Profile and Differ in Response to Atomoxetine. J Am Acad Child Adolesc Psychiatry. 2025 Jul 16:S0890-8567(25)00337-5. doi: 10.1016/j.jaac.2025.07.007. Online ahead of print. PMID 40681145
- [Derived] Arns M, Vollebregt MA, Palmer D, Spooner C, Gordon E, Kohn M, Clarke S, Elliott GR, Buitelaar JK. Electroencephalographic biomarkers as predictors of methylphenidate response in attention-deficit/hyperactivity disorder. Eur Neuropsychopharmacol. 2018 Aug;28(8):881-891. doi: 10.1016/j.euroneuro.2018.06.002. Epub 2018 Jun 22. PMID 29937325